CLINICAL TRIAL: NCT04107857
Title: Electronic Health Record-Enabled Evidence-based Smoking Cessation Quality Improvement Program
Brief Title: Electronic Health Record-Enabled Evidence-Based Smoking Cessation Quality Improvement Implementation Program
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 89276; P30CA091842 (NIH)
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Smoking Cessation: * Patients enter the program through clinic appointments or community outreach programs.
  * Patients will be given brief advice to quit smoking and referral options to receive evidence-based treatment through Missouri/Illinois Quitlines, Smokefree.TXT, or smokefree.gov dependent on the patient's preference for counseling
  * Patient can also be prescribed smoking cessation pharmacotherapy
  Interventions: Behavioral: ELEVATE enhancement to electronic health record (EHR) to improve cessation counseling offer; Behavioral: ELEVATE enhancement to electronic health record (EHR) to improve smoking cessation medication offer; Behavioral: Data Driven Feedback reports

INTERVENTIONS:
Behavioral: ELEVATE enhancement to electronic health record (EHR) to improve cessation counseling offer — * Brief advise to quit smoking
  * Referral to Missouri/Illinois Quitlines, Smokefree.TXT, or smokefree.gov
Behavioral: ELEVATE enhancement to electronic health record (EHR) to improve smoking cessation medication offer — -Nicotine replacement therapy, varenicline, bupropion, or combination therapy (not provided by study)
Behavioral: Data Driven Feedback reports — -Feedback reports will be based on data

SUMMARY:
The goal of this quality improvement program is to implement, evaluate, and sustain an evidence-based smoking cessation treatment program with a population-based approach so that all patients at the Siteman Cancer Center, Washington University, Barnes-Jewish Hospital, BJC Healthcare, and satellite locations receive assessment of smoking and all smokers receive treatment support.

ELIGIBILITY:
Inclusion Criteria:

-Patients seen at Siteman Cancer Center, Washington University, Barnes-Jewish Hospital, BJC Healthcare, or any of the satellite locations

Exclusion Criteria:

-None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age or older
Sampling Method: Non-Probability Sample
Enrollment: 1000000 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
Clinic level percentage of patients receiving brief counseling | From 6 months pre-intervention through 6 months post-intervention
Clinic level percentage of smokers offered referral to additional counseling | From 6 months pre-intervention through 6 months post-intervention
Clinic level percentage of smokers offered medication | From 6 months pre-intervention through 6 months post-intervention

SECONDARY OUTCOMES:
Clinic level percentage of patients receiving brief counseling | Estimated to be 12 months pre-intervention and 12, 24, 36, and 48 months post-intervention
Clinic level percentage of smokers offered referral to additional counseling | Estimated to be 12 months pre-intervention and 12, 24, 36, and 48 months post-intervention
Clinic level percentage of smokers offered medication | Estimated to be 12 months pre-intervention and 12, 24, 36, and 48 months post-intervention
Clinic level percentage of smokers receiving smoking assessment | Estimated to be 12 months pre-intervention and 12, 24, 36, and 48 months post-intervention
Clinic level percentage of smokers receiving cessation medication | Estimated to be 12 months pre-intervention and 12, 24, 36, and 48 months post-intervention
Number of patients who have abstained from smoking | Estimated to be 6 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Li-Shiun Chen, M.D., ScD, MPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu
- See also: Related Info — https://siteman.wustl.edu/prevention/smoking-cessation-program/